CLINICAL TRIAL: NCT04131075
Title: Microcirculatory Dysfunction in Stable Coronary Artery Disease: Relationship With Patient-focused Outcomes, Cerebral Small Vessel Disease and Depression.
Brief Title: The Cerebral-Coronary Connection (C3) Study
Acronym: C3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Salud Carlos III (Other Government)
Collaborators: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Javier Escaned, Principal Investigator, Instituto de Salud Carlos III
Other Study IDs: C3
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Ischemic Heart Disease; Microvascular Coronary Artery Disease; Depression; Endothelial Dysfunction; Inflammation
Keywords: Coronary microvascular dysfunction; Cerebral Small Vessel Diseases
MeSH Terms: conditions — Myocardial Ischemia; Depression; Inflammation; Cerebral Small Vessel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients with CAD undergoing FFR-guided revascularisation. FFR, coronary flow reserve (CFR) and the index of hyperemic microvascular resistance (HMR) will be measured with the Doppler guidewire (Combowire, Volcano - Philips corporation) under steady state hyperemia.
  Interventions: Procedure: Coronary Angiography and Multimodal Coronary Physiology Study (FFR, CFR, HMR)

INTERVENTIONS:
Procedure: Coronary Angiography and Multimodal Coronary Physiology Study (FFR, CFR, HMR) — Coronary Angiography according to clinical indication and Multimodal Coronary Physiology Study (FFR, CFR, HMR) for functional assessment of intermediate coronary lesions

SUMMARY:
This is a prospective cohort blinded study with the aim to investigate the prevalence and clinical impact of coronary microcirculatory dysfunction (CMD) in patients with ischemic heart disease, and its association with cerebral small vessel disease (CSVD) and depressive disorders. In addition, CMD and CSVD linkage to systemic inflammation and endothelial function will also be investigated.

DETAILED DESCRIPTION:
The treatment of stable CAD is largely based on a paradigm that gives epicardial coronary stenoses a central role in the generation of myocardial ischaemia. However, coronary microcirculatory dysfunction (CMD) is a major and frequently ignored cause of ischaemia that, according to retrospective studies, influences the outcomes of patients with CAD. In addition, patients with CMD may not experience symptomatic relief with myocardial revascularization or pharmacological treatment. This constitutes one of the causes of persistent angina despite successful revascularization, causing not only an impairment of the quality of life and higher consumption of healthcare resources, but potentially affective disorders like depression, which has been found to be associated with CAD and with prognosis.

It also remains largely unknown whether CMD in stable CAD is organ-specific only or rather indicative of involvement of other vital organs. While this seems to be the case in the kidney and the retina, the relationship between CMD in the heart and the brain has not been studied. Beyond classical cardiovascular risk factors linked to the development of ischemic heart disease, systemic endothelial dysfunction could constitute a link between microcirculatory involvement in both organs: the heart and the brain. Additionally, the relation between chronic inflammatory status and microvascular disease in both the heart and the brain is not known.

The principal hypotheses and sub-hypotheses are as follows:

Principal hypotheses: 1. Patients with CMD have worse prognosis compared to those ones with normal coronary microcirculation. 2. Patients with CMD have a higher prevalence of CSVD. 3. Chronic systemic inflammation status is an independent predictor of CMD and CSVD.

Sub-hypotheses: 1. The presence of CMD is associated to recurrent/persistent angina. 2. The presence of CMD is associated to higher prevalence of depressive disorders. 3. CMD and CSVD are associated to systemic endothelial dysfunction.

Primary Objectives associated to Principal hypotheses: 1. To investigate the relationship between the presence of CMD and the development of patient-focused outcomes at 1 year of follow-up. 2. To determine the prevalence of CSVD in patients with CAD with and without CMD. 3. To investigate the relationship between systemic inflammation and CMD.

Primary Objectives associated to Sub-hypotheses: 1. To determine the prevalence of persistent or recurrent angina in patients with and without CMD in whom revascularization of CAD is guided by FFR. 2. To determine the prevalence of depressive disorders in patients with and without CMD. 3. To investigate the relationship between the status of systemic endothelial function and the presence of CMD and CSVD.

Methods: Patients with CAD undergoing FFR-guided revascularisation will be prospectively enrolled. FFR, coronary flow reserve (CFR) and the index of hyperemic microvascular resistance (HMR) will be measured with the Doppler guidewire (Combowire, Volcano - Philips corporation) under steady state hyperemia (intravenous adenosine infusion, 140 mcg/Kg/min). CMD will be defined according to CFR and HMR, and will be used to classify the overall population in two groups: the study group (presence of CMD) and the control group (absence of CMD). Coronary revascularization will be decided according to result of FFR (cutoff ≤0.80).

After the procedure the patient will undergo baseline clinical assessment: • Neurological clinical assessment and Transcranial Doppler Ultrasound. • Psychiatric clinical assessment. • Stress Cardiac MRI and Cerebral MRI. • Peripheral endothelial function test with plethysmography-based device EndoPat. • Laboratory blood tests for systemic inflammation markers, platelet function and endothelial progenitor cells. • Baseline assessment of angina status by the Seattle Questionnaire of angina (SAQ).

Clinical follow-up will be performed at 1-month, 6-months and 1-year, and will include: • clinical cardiology and psychiatric assessment, assessment of angina status by the SAQ. • stress test (1-year). • peripheral endothelial function test with plethysmography-based device EndoPat (1-year). • neurological clinical assessment and Transcranial Doppler Ultrasound (1- year). • laboratory blood tests for systemic inflammation markers, platelets function and endothelial progenitor cells(1-year).

Type of blinding: Data regarding coronary microcirculation invasive assessment, neurologic and psychiatric clinical assessment, cardiac and cerebral MRI, Trans-cranial Doppler Ultrasound, laboratory blood tests, systemic endothelial function and follow-up will be collected in a blinded fashion, so that patient and the other investigators, apart from the invasive cardiology team responsible for patient enrollment and study coordination, could not access to them. Primary events rate (major adverse cardiovascular events, incidence of CSVD, systemic inflammation status, depressive disorders, recurrent angina and systemic endothelial dysfunction) will be analyzed and correlated to CMD in a blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent available.
* Age ≥ 18 years.
* Stable coronary lesions.
* Indication to FFR: ≥ 1 intermediate coronary lesion (40-80% diameter stenosis) in a principal/secondary vessel with ≥ 2 mm reference diameter.

Exclusion Criteria:

* Previous myocardial infarction in the territory of distribution of the target vessel.
* Coronary Left Main severe stenosis.
* Aortic valve stenosis (moderate or severe) .
* Severe left ventricle hypertrophy.
* Left ventricle moderate systolic dysfunction (EF < 35%).
* Contraindications to adenosine.
* Previous CABG with permeable grafts.
* Contraindication to stent implantation.
* Severe anemia.
* Coagulopathies or chronic anticoagulation.
* Platelets < 75000 o > 700.000.
* Previous stroke or intracranial hemorrhage.
* Contraindication to MRI.
* Chronic Renal Failure contraindicating gadolinium infusion during MRI: eGFR < 60 ml/min), hemodialysis, previous renal transplantation.
* Pacemaker/ Implantable Cardioverter Device with contraindication to MRI.
* Planned cardiac surgery.
* Life expectancy < 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable coronary lesions (stable coronary disease or lesions in non-culprit vessels >48 hours after acute coronary syndrome) with clinical indication to coronary angiography and intermediate coronary lesions (visual estimation) suitable for FFR-guided revascularization.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Cardiovascular Events (MACE): all-cause of death, myocardial infarction and any type of coronary revascularization | 1 month
  Clinical assessment
Incidence of Major Cardiovascular Events (MACE): all-cause of death, myocardial infarction and any type of coronary revascularization | 6 months
  Clinical assessment.
Incidence of Major Cardiovascular Events (MACE): all-cause of death, myocardial infarction and any type of coronary revascularization | 1 year
  Clinical assessment.
Prevalence of Cerebral Small Vessel Disease (CSVD). | Baseline
  Determined by Cerebral MRI, transcranial Doppler Ultrasound and clinical assessment.
Prevalence of Cerebral Small Vessel Disease (CSVD). | 1 year
  Determined by Cerebral MRI, transcranial Doppler Ultrasound and clinical assessment.

SECONDARY OUTCOMES:
Assessment of angina status by Seattle Angina Questionnaire (SAQ) | 1 month
  The SAQ (Seattle Angina Questionnaire) quantifies 5 domains measuring the impact of angina on patients' health status: Physical Limitation (9 items), Angina Stability (1 item), Angina Frequency (2 items), Treatment Satisfaction (4 items), and Quality of Life (3 items). Item responses are coded sequentially from worst to best status and range from 1 to 6 for Physical Limitation, Angina Stability, and Angina Frequency items; 1 to 5/6 for Treatment Satisfaction items; and 1 to 5 for Quality of Life items. Scores are generated for each domain and are scaled 0 to 100, with 0 denoting the worst and 100 the best possible status.
Assessment of angina status by Seattle Angina Questionnaire (SAQ) | 6 months
  The SAQ (Seattle Angina Questionnaire) quantifies 5 domains measuring the impact of angina on patients' health status: Physical Limitation (9 items), Angina Stability (1 item), Angina Frequency (2 items), Treatment Satisfaction (4 items), and Quality of Life (3 items). Item responses are coded sequentially from worst to best status and range from 1 to 6 for Physical Limitation, Angina Stability, and Angina Frequency items; 1 to 5/6 for Treatment Satisfaction items; and 1 to 5 for Quality of Life items. Scores are generated for each domain and are scaled 0 to 100, with 0 denoting the worst and 100 the best possible status.
Assessment of angina status by Seattle Angina Questionnaire (SAQ) | 1 year
  The SAQ (Seattle Angina Questionnaire) quantifies 5 domains measuring the impact of angina on patients' health status: Physical Limitation (9 items), Angina Stability (1 item), Angina Frequency (2 items), Treatment Satisfaction (4 items), and Quality of Life (3 items). Item responses are coded sequentially from worst to best status and range from 1 to 6 for Physical Limitation, Angina Stability, and Angina Frequency items; 1 to 5/6 for Treatment Satisfaction items; and 1 to 5 for Quality of Life items. Scores are generated for each domain and are scaled 0 to 100, with 0 denoting the worst and 100 the best possible status.
Prevalence of depressive and anxiety disorders, determined by clinical assessment and dedicated questionnaires. | 1 month
  An expert psychologist will perform the following assessment: i) basal depression screening (Patient Health Questionnaire [PHQ-9]); ii) Standardized Interview (International neuropsychiatric interview) iii) evaluation of the severity of depression (Montgomery-Asberg score [MDRS]); iv) anxiety symptoms detection (Hamilton anxiety rating scale [HARS]); v) assessment of baseline quality of life (The MOS 36-item Short Form Health Survey [SF-36]); vi) functional skills assessment (The Lawton Instrumental Activities of Daily Living (IADL) Scale).
Prevalence of depressive and anxiety disorders, determined by clinical assessment and dedicated questionnaires. | 6 months
  An expert psychologist will perform the following assessment: i) basal depression screening (Patient Health Questionnaire [PHQ-9]); ii) Standardized Interview (International neuropsychiatric interview) iii) evaluation of the severity of depression (Montgomery-Asberg score [MDRS]); iv) anxiety symptoms detection (Hamilton anxiety rating scale [HARS]); v) assessment of baseline quality of life (The MOS 36-item Short Form Health Survey [SF-36]); vi) functional skills assessment (The Lawton Instrumental Activities of Daily Living (IADL) Scale).
Prevalence of depressive and anxiety disorders, determined by clinical assessment and dedicated questionnaires. | 1 year
  An expert psychologist will perform the following assessment: i) basal depression screening (Patient Health Questionnaire [PHQ-9]); ii) Standardized Interview (International neuropsychiatric interview) iii) evaluation of the severity of depression (Montgomery-Asberg score [MDRS]); iv) anxiety symptoms detection (Hamilton anxiety rating scale [HARS]); v) assessment of baseline quality of life (The MOS 36-item Short Form Health Survey [SF-36]); vi) functional skills assessment (The Lawton Instrumental Activities of Daily Living (IADL) Scale).
Prevalence of systemic inflammation status, determined by laboratory blood tests. | Baseline
  Determination of blood levels of pro-inflammatory proteins (hsCRP, IL-1, IL-6, IL-18, VCAM-1 and ICAM-1) by ELISA method. Given the fact that the chronic inflammation can induce changes in the mononuclear cells phenotype, we will analyze the immune activation status (by analyzing CD4+/CD38+-T lymphocytes, CD8+/CD38+-T lymphocytes and CD8+/CD38+/HLADR+-T lymphocytes). The analysis will be performed by flow cytometry (Galios, Beckman Coulter). In addition, we will study the NRLP3 protein complex (which is involved in atherogenesis).
Prevalence of systemic inflammation status, determined by laboratory blood tests. | 1 year
  Determination of blood levels of pro-inflammatory proteins (hsCRP, IL-1, IL-6, IL-18, VCAM-1 and ICAM-1) by ELISA method. Given the fact that the chronic inflammation can induce changes in the mononuclear cells phenotype, we will analyze the immune activation status (by analyzing CD4+/CD38+-T lymphocytes, CD8+/CD38+-T lymphocytes and CD8+/CD38+/HLADR+-T lymphocytes). The analysis will be performed by flow cytometry (Galios, Beckman Coulter). In addition, we will study the NRLP3 protein complex (which is involved in atherogenesis).
Peripheral endothelial dysfunction, assessed by EndoPat. | Baseline
  Systemic endothelial dysfunction is defined as the inability of the arterial system to dilate appropriately in response to hyperaemia stimulus in order to increase blood flow according to metabolic demands. In this study, we will use the EndoPat technology that allows non-invasive evaluation of vasoreactivity by the assessment of the pulsatile arterial flow in the fingertip. We will assess changes in the flow from baseline and after inducing ischaemia by inflating a blood pressure cuff to occlude the brachial artery. Changes in endothelial measurements and in vascular tone after each occlusion of the brachial artery are a reflection of the hyperaemic vasoreactivity and endothelial function. By comparing the results during rest and ischaemia to the results obtained in the contralateral arm (which has not been subjected to ischaemia) we will obtain the index of reactive hyperaemia or EndoScore´. This Endoscore can then be used to evaluate endothelial function.
Peripheral endothelial dysfunction, assessed by EndoPat. | 1 year
  Systemic endothelial dysfunction is defined as the inability of the arterial system to dilate appropriately in response to hyperaemia stimulus in order to increase blood flow according to metabolic demands. In this study, we will use the EndoPat technology that allows non-invasive evaluation of vasoreactivity by the assessment of the pulsatile arterial flow in the fingertip. We will assess changes in the flow from baseline and after inducing ischaemia by inflating a blood pressure cuff to occlude the brachial artery. Changes in endothelial measurements and in vascular tone after each occlusion of the brachial artery are a reflection of the hyperaemic vasoreactivity and endothelial function. By comparing the results during rest and ischaemia to the results obtained in the contralateral arm (which has not been subjected to ischaemia) we will obtain the index of reactive hyperaemia or EndoScore´. This Endoscore can then be used to evaluate endothelial function.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Escaned, MD, PhD, Principal Investigator — Instituto Carlos III. Hospital Clínico San Carlos.
Locations (1):
- Hospital Clínico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mejia-Renteria H, Travieso A, Matias-Guiu JA, Yus M, Espejo-Paeres C, Finocchiaro F, Fernandez S, Gomez-Escalonilla CI, Reneses-Prieto B, Gomez-Garre MD, Delgado-Alvarez A, Bustos A, Perez de Isla L, de Diego JJG, Modrego-Martin J, Ortega-Hernandez A, Papadopoulos P, Arrazola-Garcia J, Matias-Guiu J, Escaned J. Coronary microvascular dysfunction is associated with impaired cognitive function: the Cerebral-Coronary Connection study (C3 study). Eur Heart J. 2023 Jan 7;44(2):113-125. doi: 10.1093/eurheartj/ehac521. PMID 36337036